CLINICAL TRIAL: NCT06514443
Title: Exploration of Country-specific Barriers and Facilitators for the Implementation of Physical Activity According to the EULAR Physical Activity Recommendations for People With Rheumatic Musculoskeletal Diseases in Four Different European Countries; the COPA Project
Brief Title: Barriers and Faciliators for Physical Activity in People With RMDs
Acronym: COPA
Status: Not yet recruiting | Type: Observational
Sponsor: Anne-Kathrin Rausch (Other)
Collaborators: Acibadem University (Other); Leiden University Medical Center (Other); Sorbonne University (Other)
Responsible Party: Sponsor-Investigator, Anne-Kathrin Rausch, PhD, Zurich University of Applied Sciences
Organization: Zurich University of Applied Sciences (Other)
Other Study IDs: Zurich UAS
Record Dates: First submitted 2024-07-16; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip; Rheumatoid Arthritis; Axial Spondyloarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Arthritis, Rheumatoid; Axial Spondyloarthritis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- osteoarthrits: adults with hip or knee osteoarthritis
  Interventions: Other: survey
- inflammatory arthritis: adults with rheumatoid arthritis or axial Spondyloarthritis
  Interventions: Other: survey

INTERVENTIONS:
Other: survey — survey exploring barriers and faciltiators for physical activity

SUMMARY:
The aim of this project is to systematically survey and explore barriers and facilitators for the implementation of physical activity according to the physical activity recommendations of the European Alliance of Associations for Rheumatology on country specific (e.g., environmental, cultural, organization and system) level. A questionnaire to explore/identify these barriers and facilitators in the survey, will be developed through literature search, interviews with multiple stakeholders (i.e., patients with inflammatory arthritis or osteoarthritis and physical therapists) and experts in the field in four different European countries (i.e., Turkey, Switzerland, the Netherlands and France).

Additionally, in Switzerland only, the Inflammatory Arthritis Facilitators and Barriers to Physical Activity (IFAB) Questionnaire which was developed to determine the factors on personal level, will be translated into the German language. Aim is to evaluate the validity and reliability of the IFAB Questionnaire in the German-speaking population with axial Spondyloarthrits, and to perform a cultural adaptation if necessary at the same time.

ELIGIBILITY:
Inclusion Criteria:

* adults being 18years or older
* diagnosis of osteoarthritis, rheumatoid arthritis or axial Spondyloarthritis
* the cognitive and linguistic competencies to answer the survey

Exclusion Criteria:

* having a rheumatological or musculoskeletal disease other than described
* any communication problems

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: people with osteoarthritis, rheumatoid arthritis or axial Spondyloarthritis living in Turkey, the Netherlands, France or Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-12-23 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
barriers and facilitators for physical activity | September-December 2024
  factors on social, envirionmental or system level impacting the physial activity behaviour

SECONDARY OUTCOMES:
reliability of the IFAB | September-December 2024
  ONLY Swiss participants with axSpA
validity of the IFAB | September-December 2024
  ONLY Swiss participants with axSpA